CLINICAL TRIAL: NCT02855346
Title: A Phase 1, Randomized, Double-Blind Pharmacokinetic and Safety Study of Dapivirine/Levonorgestrel Vaginal Rings
Brief Title: PK and Safety Study of Vaginal Rings Containing Dapivirine and Levonorgestrel
Acronym: DAP/LNG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MTN-030/IPM 041; 5UM1 A1068633 (Other Grant/Funding Number: Division of AIDS, US National Institute of Allergy and Infectious Diseases US Eunice Kennedy Shriver National Institute)
Record Dates: First submitted 2016-06-21; First posted 2016-08-04 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: HIV Prevention
MeSH Terms: interventions — Dapivirine; Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 200 mg of DPV (Experimental): Each participant will receive a VR containing either 200 mg DPV or 200 mg DPV + 320 mg LNG. Participants will be randomized in a 1:1 ratio. The VR should be worn for approximately 14 consecutive days +/-1 day. The ring will be removed by the participant (or clinician/designee, if necessary) at the Product Use End Visit (PUEV)/Early Termination Visit. The participant will be followed for approximately 2 days following VR removal
  Interventions: Combination Product: 200 mg of DPV + 320 mg LNG
- 200 mg of DPV + 320 mg LNG (Experimental): Each participant will receive a VR containing either 200 mg DPV or 200 mg DPV + 320 mg LNG. Participants will be randomized in a 1:1 ratio. The VR should be worn for approximately 14 consecutive days +/-1 day. The ring will be removed by the participant (or clinician/designee, if necessary) at the Product Use End Visit (PUEV)/Early Termination Visit. The participant will be followed for approximately 2 days following VR removal
  Interventions: Combination Product: 200 mg of DPV

INTERVENTIONS:
Combination Product: 200 mg of DPV + 320 mg LNG — DPV VR, containing 200 mg DPV
  Other Names: Dapivirine
  Arms: 200 mg of DPV
Combination Product: 200 mg of DPV — DPV-LNG VR, containing 200 mg of DPV + 320 mg LNG
  Other Names: Dapivirine/Levonorgestrel
  Arms: 200 mg of DPV + 320 mg LNG

SUMMARY:
PK and Safety Study of Vaginal Ring Containing Dapivirine and Levonorgestrel

DETAILED DESCRIPTION:
A Phase 1, Randomized, Double-Blind Pharmacokinetic and Safety Study of Dapivirine/Levonorgestrel

ELIGIBILITY:
Inclusion Criteria:

* Healthy women

Exclusion Criteria:

* HIV infected women

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
Dapivirine and levonorgestrel concentrations in blood and Vaginal fluid | 14 days
  To characterize the local and systemic pharmacokinetics of one dapivirine vaginal ring formulation and one dapivirine-levonorgestrel vaginal ring formulations used continuously for 14 days

SECONDARY OUTCOMES:
Grade 2 or higher Genitourinary adverse event and Grade 3 or higher adverse event as defined by DAIDS | 14 days
  To evaluate the safety of one dapivirine vaginal ring formulation and one dapivirine-levonorgestrel vaginal ring formulations used continuously for 14 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama Hospital, Birmingham, Alabama
  - Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Friedland BA, Gundacker H, Achilles SL, Chen BA, Hoesley C, Richardson BA, Kelly CW, Piper J, Johnson S, Devlin B, Steytler J, Kleinbeck K, Dangi B, Friend C, Song M, Mensch B, van der Straten A, Jacobson C, Hendrix CW, Brown J, Blithe D, Hiller SL; MTN-030/IPM 041 and MTN-044/IPM 053/CCN019 Protocol Teams for the Microbicide Trials Network and the Contraceptive Clinical Trials Network. Acceptability of a dapivirine levonorgestrel vaginal ring in two Phase 1 trials (MTN-030/IPM 041 and MTN-044/IPM 053/CCN019): Implications for multipurpose prevention technology development. PLoS One. 2025 Jan 14;20(1):e0312957. doi: 10.1371/journal.pone.0312957. eCollection 2025. PMID 39808648